CLINICAL TRIAL: NCT06116825
Title: The Effect of Brushing With Fluoride Toothpaste on Dental Plague Control for Elementary School Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KMUHIRB-SV(I)-20220008
Record Dates: First submitted 2023-10-31; First posted 2023-11-03 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2022-05

CONDITIONS: Healthy
Keywords: children; Health Education; brushing technique; dental plaque
MeSH Terms: conditions — Health Education; Dental Plaque

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experiment group (Experimental): In the experimental group, students from grades three to six in four primary schools in Chiayi County participated. Participating school children are taught the correct method of brushing their teeth, and flossing is also taught in the upper grades. The experimental group used toothpaste containing 1,450 ppm fluoride and asked students to use it at least twice a day, one of which was to clean their teeth before bed. During the pre-test and 4-week post-test, the plaque control index (Plaque Control Record; PCR) was checked and a self-administered questionnaire was filled out.
  Interventions: Other: 1450ppm Fluoride toothpaste
- Control group (Active Comparator): In the control group, students from grades three to six in four primary schools in Chiayi County participated. All participating children receive instruction on proper tooth brushing techniques, with flossing included in higher grades. Schoolchildren in the control group were given toothpaste containing 1,000 ppm fluoride and were asked to use it at least twice a day, including once to clean their teeth before bed. During the pre-test and 4-week post-test, the plaque control index (Plaque Control Record; PCR) was checked and a self-administered questionnaire was filled out.
  Interventions: Other: 1000Pppm Fluoride toothpaste

INTERVENTIONS:
Other: 1450ppm Fluoride toothpaste — 1450ppm Fluoride toothpaste
  Arms: Experiment group
Other: 1000Pppm Fluoride toothpaste — 1000Pppm Fluoride toothpaste
  Arms: Control group

SUMMARY:
The purpose of this study is to evaluate the effect of correct tooth cleaning and use of fluoride toothpaste after school lunch and before going to bed on primary school children's plaque reduction and tooth cleaning skills.

DETAILED DESCRIPTION:
Taking the school as a unit, the participants are children in grades three to six of elementary schools under the jurisdiction of Chiayi County, with a total expected sample size of 400 people.

Through class teaching, the Shelley method of brushing teeth is taught, and flossing instruction is added to senior grades to improve students' teeth cleaning skills. They also use fluoride toothpaste with a concentration of more than 1000PPM to clean teeth after lunch at school and before going home to go to bed. School children were tested for plaque before and after using fluoride toothpaste, collected plaque control index, filled out a self-administered tooth cleaning skills and self-efficacy questionnaire, and tracked changes in the six weeks after use.

Professional dentists and researchers will go to school to conduct dental plaque testing and fill out the first questionnaire for students. They will also use fluoride toothpaste after lunch at school and before going home to go to bed. Together with correct tooth cleaning methods, at 6 weeks Afterwards, the dental plaque test will be carried out again and the second questionnaire will be filled out. Each filling in of the questionnaire will take about ten minutes.

ELIGIBILITY:
Inclusion Criteria:

* Chiayi County has jurisdiction over elementary school students in grades three to six

Exclusion Criteria:

- 1. Students with disability certificates. 2. School children with congenital serious oral diseases (such as cleft lip and palate).

3. Children who are unable to operate the Bates tooth brushing method (such as students who are still unable to complete the operation after being guided by teachers and researchers).

Ages: 9 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 400 (Actual)
Dates: Start 2022-10-20 (Actual); Primary Completion 2022-12-27 (Actual); Study Completion 2022-12-27 (Actual)

PRIMARY OUTCOMES:
Plaque Control Record (PCR) | Change from Baseline PCR at 6-week after intervention
  The Plaque Control Record is a very simple percentage or score of the total amount of bacteria present in your mouth.
  A tooth has 6 surfaces at the gum line being; the lingual side (distal, middle, mesial) and buccal side (distal, middle, mesial). For each patient, PCR will measured each teeth.

SECONDARY OUTCOMES:
Teeth cleaning skill | Change from Baseline at 6-week after intervention
  Teeth cleaning skill is a questionnaire scale. Total of 5 items ex. What method do I usually use to brush my teeth?
Self-efficacy | Change from Baseline at 6-week after intervention
  Self-efficacy is a questionnaire scale. Total of 2 items ex.I am confident that I can brush my teeth clean

CONTACTS AND LOCATIONS:
Overall Officials: HSIAO-LING HUANG, Dr.PH, Principal Investigator — Kaohsiung Medical University, College of Dental Medicine, Department of Oral Hygiene
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Taiwan